CLINICAL TRIAL: NCT00851045
Title: A Randomized, Double-Blind, Phase II Trial of CT-322 (BMS-844203) Plus Irinotecan, 5-FU and Leucovorin (FOLFIRI) Versus Bevacizumab Plus FOLFIRI as Second-Line Treatment for Metastatic Colorectal Cancer
Brief Title: Ph II Trial of a Novel Anti-angiogenic Agent in Combination With Chemotherapy for the Second-line Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA196-004; EUDRACT # 2008-006561-89
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin; CT-322; Bevacizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Irinotecan/5-Fluorouracil (bolus)/5-Fluorouracil (infusional)/Leucovorin calcium/CT-322
  Interventions: Drug: Irinotecan; Drug: 5-Fluorouracil (bolus); Drug: 5-Fluorouracil (infusional); Drug: Leucovorin calcium; Drug: CT-322
- Arm 2 (Active Comparator): Irinotecan/5-Fluorouracil(bolus)/5-Fluorouracil(infusional)/Leucovorin calcium /Bevacizumab/Bevacizumab Placebo(saline solution)
  Interventions: Drug: Irinotecan; Drug: 5-Fluorouracil (bolus); Drug: 5-Fluorouracil (infusional); Drug: Leucovorin calcium; Drug: Bevacizumab; Drug: Bevacizumab Placebo (saline solution)

INTERVENTIONS:
Drug: Irinotecan — Solution, IV, 180 mg/m2, Q14 days, Until PD
  Other Names: Camptosar
Drug: 5-Fluorouracil (bolus) — Solution, IV, 400 mg/m2, Q14 days, Until PD
Drug: 5-Fluorouracil (infusional) — Solution, IV, 2400 mg/m2, Q14 days, Until PD
Drug: Leucovorin calcium — Solution, IV, 400 mg/m2, Q14 days, Until PD
Drug: CT-322 — Solution, IV, 2 mg/kg, Q7 days, Until PD
  Other Names: BMS-844203
  Arms: Arm 1
Drug: Bevacizumab — Solutions, IV, 5 mg/kg, Q14 days, Until PD
  Other Names: Avastin
  Arms: Arm 2
Drug: Bevacizumab Placebo (saline solution) — Solution, IV, 0 mg/kg, On day 8 of a 2-week cycle, Until PD
  Other Names: Saline Solution
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the efficacy of CT-322 comparative to bevacizumab, both in combination with irinotecan, 5-FU and leucovorin in the second-line treatment of subject with metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status (PS) ≤1
* Histologically or cytologically confirmed, unresectable metastatic colorectal cancer
* Measurable disease by RECIST guidelines
* Evidence of disease progression following first-line therapy with a fluoropyrimidine, oxaliplatin, and bevacizumab (≤ 8 weeks since last dose)
* Available paraffin embedded tumor tissue
* Willing to give a whole blood sample for the study of proteins and genetic polymorphisms

Exclusion Criteria:

* Less than 28 days elapsed since major surgery at time of randomization
* Known CNS metastases
* Excessive risk of bleeding (including use of therapeutic anticoagulation other than low dose aspirin) and history of thrombotic or embolic cerebrovascular accident
* Uncontrolled hypertension
* Clinically significant cardiovascular disease
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Serious non-healing wound, active peptic ulcer, non-healing bone fracture, or bleeding skin metastasis
* Known HIV Positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival based on tumor assessments (CT/MRI) | Every 6 weeks until documented progressive disease, initiation fo subsequent therapy for colorectal cancer, or withdrawal of consent

SECONDARY OUTCOMES:
Overall survival (OS), defined as the time the subject is randomized until death, in each arm | every 12 weeks
Objective tumor response rate (ORR), defined as the proportion of randomized subjects in each arm whose best response is CR (complete response) or PR (partial response) using RECIST guidelines as determined by the site investigator | every 6 weeks
Safety in the CT-322 plus irinotecan, 5-FU and leucovorin arm as measured by incidence of serious and non-serious adverse events, significant laboratory evaluations and significant physical examination findings in subjects | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (12):
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Compassionate Cancer Care Medical Group Inc, Fountain Valley, California
  - Compassionate Cancer Care Medical Group, Inc, Riverside, California
  - Sharp Memorial Hospital, San Diego, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Midwest Center For Hematology/Oncology, Joliet, Illinois
  - Cancer Center Of Kansas, Wichita, Kansas
  - Gurtler, Jayne, Metairie, Louisiana
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
  - Pharma Resource, East Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University Of Texas M.D. Anderson Cancer Center, Houston, Texas
- Argentina (2):
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Local Institution, Terni, Italy

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx